CLINICAL TRIAL: NCT02463201
Title: Obstructive Sleep Apnea in Obese Children and Teenagers - Occurrence and Importance of Intervention
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Collaborators: Holbaek Sygehus (Other)
Responsible Party: Sponsor
Other Study IDs: SJ-404
Record Dates: First submitted 2015-06-02; First posted 2015-06-04 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Sleep Apnea, Obstructive; Pediatric Obesity
Keywords: Sleep Apnea, Obstructive; Pediatric Obesity
MeSH Terms: conditions — Sleep Apnea, Obstructive; Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Obese children and adolescents: Attending a weightloss programme, that consist of lifestyle counseling, dietary restriction and exercise. The prevalence of obstructive sleep apnea (OSA) will be investigated in group. Children diagnosed with OSA will be followed to investigate if weight loss changes the condition.
  Interventions: Behavioral: Weight loss

INTERVENTIONS:
Behavioral: Weight loss

SUMMARY:
The prevalence of childhood obesity has increased at an alarming rate over the last decades, both globally and in Denmark. There are a number of serious sequelae related to obesity, such as hypertension, hypercholesterolemia, fatty liver and prediabetes. Obesity is found to be a risk factor for obstructive sleep apnea (OSA). OSA in childhood is known to be associated with cardiovascular complications, neurocognitive problems and reduced quality of life. The correlation between obesity and OSA is still poorly understood. Early detection and intervention is of great importance as the health consequences related to OSA as well as obesity are severe. Adenotonsillectomy is recommended as first-line therapy in children with OSA. However, only around 25% of obese children benefit from this treatment compared to around 75% of normal-weight children suggesting that there might be other structural factors predisposing to OSA in obese children.

In this study the investigators aim to clarify the impact of obesity in the development of OSA. The prevalence of OSA in obese children will be investigated. Furthermore the purpose is to assess the effect of weight loss on OSA.

ELIGIBILITY:
Inclusion Criteria:

* Age: 7-18 years
* BMI > 90th percentile for age and gender

Exclusion Criteria:

* Neuromuscular disorders
* Craniofacial syndromes / malformations
* Laryngeal and tracheal malformations

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The cohort consists of children attending the Childrens Obesity Clinic in Holbaek.
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2015-04; Primary Completion 2018-02 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Change in obstructive sleep apnea (OSA) | One year
  OSA will be diagnosed by cardiorespiratory measurement. The examination will be repeated after weight loss.

CONTACTS AND LOCATIONS:
Overall Officials: Ida Andersen, MD, Principal Investigator
Locations (2):
- Denmark (2):
  - Holbaek Sygehus, Holbæk, Danmark
  - Zealand University Hospital, Køge, Danmark

REFERENCES:
- [Derived] Orntoft M, Andersen IG, Homoe P. Agreement between manual and automatic analyses of home sleep examinations in pediatric obstructive sleep apnea. J Comp Eff Res. 2019 Jun;8(8):623-631. doi: 10.2217/cer-2018-0093. Epub 2019 May 24. PMID 31122047